CLINICAL TRIAL: NCT07358325
Title: Effectiveness of a Video-Based Educational Intervention Compared With In-Person Education on Psychosocial and Functional Outcomes in Patients Undergoing Arthroscopic Partial Meniscectomy: A Noninferiority Randomized Controlled Trial
Brief Title: Video-Based Education Versus In-Person Education in Patients Undergoing Arthroscopic Partial Meniscectomy
Acronym: NI-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CLF23/05
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Partial Meniscectomy; Knee Arthroscopic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based group (Experimental): Subjects assigned to this group will be asked to watch educational video within 5 days before surgery and to performe exercises shown in the video during the 2 weeks after surgery.
  Interventions: Behavioral: Video-based education
- Control group (Active Comparator): Subjects assigned to this group will be instructed in-person by a physiotherapist on educational advice and exercises to perform during the 2 weeks after surgery.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Video-based education — The video-based education was sent to patients within 5-day before surgery and consists of instructions to follow after surgery on wight-baring on the operated limb, advice to reduce swelling and movements tallowed to be performed. Exercises to perform in the 2 weeks after surgery are shown.
  Arms: Video-based group
Behavioral: Usual Care — Immediately after the surgery in day-hospital setting, a physiotherapist provided in-person instructions to patients assigned to control group. Instructions consists of the same educational content of the video-based group and the same exercises to perform in 2-weeks after surgery are shown and provided on a written spreadsheet.
  Arms: Control group

SUMMARY:
The primary aim of the study is to investigate whether video-based education and exercise-program is non-inferior to in-person instructions in improving pain-related self-efficacy in patients undergoing arthroscopic partial meniscectomy in a day-hospital setting. Secondary aims are to explore the potential superiority of the video-based program compared to in-person instructions in reducing disability and kinesiophobia in the same patient population.

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled for arthroscopic partial meniscectomy (medial or lateral meniscus) performed in a day-hospital setting.
* Traumatic or degenerative meniscal tears.
* Treatment at the Hip and Knee Orthopedic Unit of the Humanitas Clinical Institute.
* Age ≥ 18 years.
* Access to adequate video support.
* Sufficient proficiency in the Italian language.

Exclusion Criteria

* Previous surgery on either knee within the past 5 years.
* Significant postoperative hematoma requiring aspiration.
* Neurological conditions potentially affecting functional or motor recovery.
* Musculoskeletal conditions potentially affecting functional or motor recovery.
* Rheumatologic conditions potentially affecting functional or motor recovery.
* Internal medicine conditions potentially affecting functional or motor recovery.
* Oncological conditions potentially affecting functional or motor recovery.
* Cognitive or psychiatric disorders (Mini-Mental State Examination ≤ 21).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain Self-Efficacy Questionnaire (PSEQ) | From enrolment to the 6 weeks after surgery
  The PSEQ assesses patients' confidence in performing daily activities despite pain, with score ranging from 0 to 60 and higher scores indicating greater pain-related self-efficacy.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From enrolment to the 3 weeks after surgery
  The WOMAC evaluates knee pain, stiffness, and physical function, with score ranging from 0 to 96 and higher scores reflecting greater pain and functional impairment.
Tampa Scale of Kinesiophobia (TSK) | From enrolment to the 3 weeks after surgery
  The TSK measures fear of movement and re-injury related to pain, with score ranging from 17 to 68 and higher scores indicating greater levels of kinesiophobia.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From enrolment to the 6 weeks after surgery
  The WOMAC evaluates knee pain, stiffness, and physical function, with score ranging from 0 to 96 and higher scores reflecting greater pain and functional impairment.
Tampa Scale of Kinesiophobia (TSK) | From enrolment to the 6 weeks after surgery
  The TSK measures fear of movement and re-injury related to pain, with score ranging from 17 to 68 and higher scores indicating greater levels of kinesiophobia.
Pain Self-Efficacy Questionnaire (PSEQ) | From enrolment to the 3 weeks after surgery
  The PSEQ assesses patients' confidence in performing daily activities despite pain, with score ranging from 0 to 60 and higher scores indicating greater pain-related self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed in this study are available on request from the corresponding author.